CLINICAL TRIAL: NCT00272441
Title: Prevention of Early Asthma in Kids (PEAK)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Childhood Asthma Research and Education Network (Network)
Model: Crossover | Purpose: Treatment
Other Study IDs: 350; NCT00000622 (obsolete NCT alias)
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

INTERVENTIONS:
Drug: inhaled corticosteroids

SUMMARY:
To evaluate current and novel therapies and management strategies for children with asthma. The emphasis is on clinical trials that help identify optimal therapy for children with different asthma phenotypes, genotypes, and ethnic backgrounds and children at different developmental stages.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a complex disease that often starts early in life. Exacerbations can be triggered by a number of agents such as allergens, respiratory infections, environmental tobacco smoke and pollutants, drugs, chemicals, exercise, cold air, infections and strong emotion making asthma therapy difficult and sometimes complicated. Multiple medications are often required to treat symptoms (bronchodilator agents such as beta-2 adrenergic agonists, theophylline, and anticholinergics), as well the underlying disease process (anti-inflammatory agents such as inhaled and systemic corticosteroids, cromolyn sodium and nedocromil; and leukotriene modifiers).

The prevalence of asthma is increasing in all age groups, but most particularly in children under the age of 18 years. In 1992, the prevalence of self-reported asthma among persons under 18 years of age was 7.2 percent, compared to 5.1 percent among all persons. The most rapid increase in asthma has occurred in children under 5 years old, with rates increasing over 160 percent over the past 15 years. Among all ages, over 450,000 hospitalizations, 5,000 deaths, and more than 100 million days of restricted activity are due to asthma every year. Yet the burden of asthma disproportionately affects children. For example, asthma hospitalization rates are highest among persons age 0-4 years, and have increased over 28 percent in the last 15 years; mortality rates increased faster among those aged 5 to-12 years than among those age 15-34 years and neither changes in disease coding nor improved recognition of asthma fully explain these increases. Nearly one third of children restrict their activities due to asthma, including participation in physical education and sports.

Despite major advances in understanding the etiology and pathophysiology of asthma and the development of new therapeutic modalities to control symptoms and prevent exacerbations, effective therapies are not widely used in the pediatric health care community. Further, the long term effects and side effects of asthma medications in children, especially children under the age of 12 years, are not well understood. Much remains to be learned about the impact of asthma therapy at different ages and at different points in the natural history of the asthma in altering the progression, chronicity, or severity of the disease.

There is an urgent need to rapidly evaluate new and existing therapeutic approaches for children with asthma, and to disseminate the findings to health care professionals, patients and the public. There are several reasons why a pediatric asthma clinical research network will accelerate clinical research and meet this need. The highly variable and sometimes complicated clinical manifestations of asthma often make it difficult to accumulate a large number of comparable patients in one center. Further, uniformity in treatment protocols may reduce the number of patients needed at each clinical center. Also, the network mechanism will help pool the necessary clinical expertise and administrative resources to facilitate the conduct of multiple and novel therapeutic trials in a timely, efficient manner. This, in turn, would promote rapid dissemination of research findings to health care professionals.

DESIGN NARRATIVE:

Prevention of Early Asthma in Kids (PEAK) began recruitment in January 2001 and evaluated whether administering inhaled corticosteroids to 24-48 month old children at risk of developing asthma prevented the development of persistent asthma. All subjects were expected to be randomized prior to December 2001 with study completion by September 2004. The study was a double blind, randomized, placebo controlled, parallel comparison of inhaled fluticasone to placebo. There was a four week run-in period to qualify and characterize children. A total of 285 children were randomized to one of two treatment groups; one receiving active treatment, the other placebo. The study was based on a continuous treatment schedule for a period of twenty-four months, followed by an observation period of one year during which the main outcomes were assessed. The primary outcome measure was the number of asthma-free days. Secondary outcomes included number of exacerbations, use of asthma medications, and lung function. There were three specific objectives of the study: 1) To assess if chronic therapy with inhaled corticosteroids initiated in children four years or less at high risk of developing asthma can prevent the development of significant asthma at four to six years of age, 2) To determine if asthma therapy as described above can prevent both losses in lung function and the development of bronchial hyperresponsiveness (BHR) associated with early onset asthma, and 3) To assess potential side effects that may be associated with long term use of inhaled steroids in early life. PEAK study outcomes were presented at the 2005 annual meetings of the American Academy of Allergy, Asthma, and Immunology and the American Thoracic Society. A manuscript has been submitted for publication by the New England Journal of Medicine.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Asthmatic children from birth to 18 years. Emphasis is placed on infants and young children through 5 years of age.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2001-01; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vernon Chinchilli — Milton S. Hershey Medical Center; Robert Lemanske — University of Wisconsin, Madison; Fernando Martinez — University of Arizona; Robert Strunk — Washington University School of Medicine; Stanley Szefler — National Jewish Health; Robert Zeiger — University of California, San Diego

REFERENCES:
- [Result] Guilbert TW, Morgan WJ, Zeiger RS, Mauger DT, Boehmer SJ, Szefler SJ, Bacharier LB, Lemanske RF Jr, Strunk RC, Allen DB, Bloomberg GR, Heldt G, Krawiec M, Larsen G, Liu AH, Chinchilli VM, Sorkness CA, Taussig LM, Martinez FD. Long-term inhaled corticosteroids in preschool children at high risk for asthma. N Engl J Med. 2006 May 11;354(19):1985-97. doi: 10.1056/NEJMoa051378. PMID 16687711
- [Derived] Bacharier LB, Phillips BR, Zeiger RS, Szefler SJ, Martinez FD, Lemanske RF Jr, Sorkness CA, Bloomberg GR, Morgan WJ, Paul IM, Guilbert T, Krawiec M, Covar R, Larsen G, Mellon M, Moss MH, Chinchilli VM, Taussig LM, Strunk RC; CARE Network. Episodic use of an inhaled corticosteroid or leukotriene receptor antagonist in preschool children with moderate-to-severe intermittent wheezing. J Allergy Clin Immunol. 2008 Dec;122(6):1127-1135.e8. doi: 10.1016/j.jaci.2008.09.029. Epub 2008 Oct 30. PMID 18973936